CLINICAL TRIAL: NCT01011400
Title: Measurements of the Fetal Clitoris by 2D Ultrasound
Brief Title: Ultrasonic Measurements of the Clitoris in Fetuses
Status: Withdrawn | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 121-09
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Ambiguous Genitalia
Keywords: clitoris
MeSH Terms: conditions — Disorders of Sex Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Abnormal enlargement of the clitoris in fetal life may be a sign for different pathologies. To the investigators knowledge there is no published nomogram of the clitoris size through gestation and it's assessment is usually subjective. The purpose of this study is to create a nomogram of clitorial size through gestation by measuring its size in fetuses of different age in the second and third trimester.

ELIGIBILITY:
Inclusion Criteria:

* well dated pregnancy
* singleton pregnancy
* female fetus
* appropriate for gestational age

Exclusion Criteria:

* small for gestational age
* other fetal anomalies
* maternal conditions that can cause exposure of the fetus to high androgen environment

Ages: 14 Weeks to 37 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pregnant women with a female fetus in the second or 3 ed trimester
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel